CLINICAL TRIAL: NCT06427109
Title: Omega-3 Fatty Acid Intake and Risk of Colorectal Adenoma
Brief Title: Omega-3 Fatty Acid and Colorectal Adenoma
Status: Completed | Type: Observational
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Sang Hoon Kim, Assistant Professor, Chung-Ang University
Other Study IDs: O3FA
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Neoplasms; Adenoma Colon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Dietary intake of omega-3 fatty acid — Participants were stratified into omega-3 consumption quartiles to assess colorectal adenoma incidence trends

SUMMARY:
Patients aged >40 years who underwent elective colonoscopies were recruited from ten institutions. Patients with a history of colorectal cancer or long-term dietary interventions were excluded. Participants completed a food frequency questionnaire (FFQ) prior to endoscopy. FFQ data were analyzed using energy-, age-, sex-, and body mass index-adjusted models; the dietary supplemental omega-3 intake was analyzed separately. Colonoscopy outcome data, including the adenoma number, pathology, and location, were collected. Participants were stratified into omega-3 consumption quartiles to assess colorectal adenoma incidence trends using P for trend analysis.

ELIGIBILITY:
Inclusion Criteria:

* all patients aged more than 40 years of age, scheduled for elective colonoscopy.

Exclusion Criteria:

* inflammatory bowel diseases
* history of colorectal neoplasms
* prior gastrointestinal surgery
* substance abuse including alcohol
* an inability to complete the survey due to emergency endoscopy
* cognitive impairments and those undergoing significant dietary modifications

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multi-center, nationwide cohort in Korea
Sampling Method: Non-Probability Sample
Enrollment: 798 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Colorectal adenoma | at the completion of the colonoscopy procedure
  among groups with different omega-3 intake levels

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jeong Lim, Principal Investigator — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi Province, South Korea

IPD SHARING:
Plan to Share IPD: No